CLINICAL TRIAL: NCT00109096
Title: A Randomized, Double-Blind Phase 2 Study of Two Doses of Pemetrexed in the Treatment of Platinum-Resistant, Epithelial Ovarian or Primary Peritoneal Cancer
Brief Title: Study of Pemetrexed in the Treatment of Patients With Ovarian Cancer Who Have Failed Prior Platinum-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9710; H3E-MC-JMHF
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Ovarian Neoplasms; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed

SUMMARY:
The purposes of this study are to determine: - whether standard or higher doses of pemetrexed should be given to patients with ovarian or primary peritoneal cancer that has recurred; - the safety and side effects of standard and higher doses of pemetrexed given to patients with ovarian or primary peritoneal cancer that has recurred; - whether standard or higher doses of pemetrexed can help patients with ovarian or primary peritoneal cancer that has recurred.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have been diagnosed with ovarian or primary peritoneal cancer
* Patient must have had 1 or 2 prior platinum-based chemotherapeutic regimens.
* Patient must have adequate health status.
* Patient compliance and geographic proximity that allow for adequate follow up is required.
* Signed informed consent from the patient or legal representative is required.

Exclusion Criteria:

* Patient is pregnant or breast-feeding
* Patient has received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Patient has previously participated in another study investigating pemetrexed.
* Patient is unable or unwilling to take folic acid, vitamin B12 supplementation, and corticosteroids.
* Patient cannot be taking nonsteroidal anti-inflammatory drugs around the time of administration of study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-06; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To assess the anti-tumor activity, as measured by tumor response rate (proportion of patients with complete or partial response, of 500 mg/m2 vs. 900 mg/m2 of pemetrexed therapy administered every 21 days

SECONDARY OUTCOMES:
Time to response
Duration of response
Time to objective progressive disease (TtPD)
Time to treatment failure (TtTF)
Objective PFS
OS
To assess safety and toxicity profile of two doses of pemetrexed in patients with ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- Germany (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Homburg/Saar
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Magdeburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolfsburg
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaén
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newcastle upon Tyne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sutton

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com